CLINICAL TRIAL: NCT02529423
Title: Multi-country cOllaborative Project on the rOle of Diet, FOod-related Behaviour, and Obesity in the Prevention of Depression (MoodFOOD)
Brief Title: Multi-country Project on the Role of Diet, Food-related Behavior, and Obesity in the Prevention of Depression
Acronym: MoodFOOD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Balearic Islands (Other)
Collaborators: VU University of Amsterdam (Other); University of Exeter (Other); University of Leipzig (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: FP7KKBE20132101
Record Dates: First submitted 2015-08-02; First posted 2015-08-20 (Estimated); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Depression
Keywords: food intake; food-related behaviour; obesity; socioeconomic environment; depression; nutritional strategies
MeSH Terms: conditions — Depression; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo
- Multi-nutrient supplement (Experimental): Multi-nutrient supplement
  Interventions: Dietary Supplement: Multi-nutrient supplement
- Placebo + Behavioral Activation (Experimental): Placebo + Behavioral Activation
  Interventions: Behavioral: Behavioral Activation; Other: Placebo
- Multi-nutrient + Behavioral Activation (Experimental): Multi-nutrient + Behavioral Activation
  Interventions: Dietary Supplement: Multi-nutrient supplement; Behavioral: Behavioral Activation

INTERVENTIONS:
Dietary Supplement: Multi-nutrient supplement — * Omega 3 fatty acids
  * Folic acid
  * Calcium
  * Selenium
  * Vitamin D3
  Arms: Multi-nutrient + Behavioral Activation; Multi-nutrient supplement
Behavioral: Behavioral Activation — 21 sessions (15 individual sessions and 6 group sessions) The intervention will include detailed analysis of each individual's behavior to determine idiosyncratic triggers and functions of unhelpful (e.g., mood-related snacking) and helpful food-related behavior, thereby, to reinforce helpful behaviors and to implement effective alternatives to unhelpful behaviors, building on behavioural approaches proven effective in depression.
  Arms: Multi-nutrient + Behavioral Activation; Placebo + Behavioral Activation
Other: Placebo — Placebo pills identical in look and taste but including no active ingredients
  Arms: Placebo; Placebo + Behavioral Activation

SUMMARY:
The study examines the feasibility and effectiveness of two different nutritional strategies (multi-nutrient supplement and food-related behavioural change) to prevent depression in high-risk overweight European Union citizens. Interventions will last 12 months. Design is a two-by-two factorial randomized controlled prevention trial with four intervention groups:

1. Control group (daily placebo supplements)
2. Multi-nutrient supplementation group (daily multi-nutrient supplement)
3. Food-related behavioural change group (food-related behavioural activation focusing on improving overall diet + placebo supplements)
4. Multi-nutrient supplementation + food-related behavioural activation group (daily multi-nutrient supplement + food-related behavioural activation focusing on improving overall diet).

Follow-up assessment will be conducted at 3, 6, and 12 months for primary and secondary endpoints, and during intervention for compliance, adverse events and mediating variables.Data will first be analyzed according to the intention-to-treat principle, using (mixed model) analysis of covariance with primary and secondary endpoints, testing for the effects of the two nutritional strategies separately as well as combined.

DETAILED DESCRIPTION:
Research has shown that nutrition may be an important way to promote mood and health, but so far researchers do not know which aspects of nutrition and behaviour are most important. The study is collaboration between the United Kingdom, Germany, Netherlands and Spain, funded by the European Commission. The trial compares different nutritional and lifestyle strategies that might promote mood and health in people who are overweight. For this purpose the design is a two-by-two factorial randomized controlled prevention trial with two intervention conditions: a multi-nutrient supplement and a food-related behavioural change (FBC) intervention. A total of four intervention groups are created: control condition (placebo, no FBC intervention), placebo with FBC intervention, multinutrient supplement with no FBC intervention, multi-nutrient supplement with FBC intervention.Recruitment: 1000 subjects will be recruited at four study sites in different EU countries (United Kingdom, Germany, Netherlands and Spain). Participants will be randomized with equal probability to the four intervention arms using a blind computerised randomization procedure.The multinutrient supplement and the placebo needs to taken every day during one year. The multinutrient supplement pill will contain omega 3 fatty acids, vitamin D, folic acid, selenium and calcium. FBC will consist of 21 behavioral activation sessions to adopt healthy diet behaviours that are known to explain the association between food intake and depression.

Follow-up assessment will be conducted by researchers unaware of the randomization status at 3, 6, and 12 months for primary and secondary outcomes. Data will first be analyzed according to the intention-to-treat principle, using (mixed model) analysis of covariance with primary and secondary endpoints, testing for the effects of the two nutritional strategies separately as well as combined (following the 2x2 factorial design of the trial). Per-protocol analyses and mediation analyses will be conducted to examine to what extent compliance and potential mediating mechanisms explain the impact on the primary and secondary endpoints. Data collection at the different sites will be conducted according to the strictest European code of ethics and conduct as well as codes for Good Clinical Practice, and local/national and international laws and regulations, including the Declaration of Helsinki. In a random subsample of trial participants (n=50 per intervention arm) blood samples will be collected at baseline, and after 3 and 12 months to measure blood levels of the nutrients provided with the multi-nutrient supplement.

ELIGIBILITY:
Inclusion Criteria:

* Age 18- 75 years
* Body Mass Index 25-40
* PHQ-9 score ≥ 5

Exclusion Criteria:

* Current (in past 6 months) clinical Major Depressive Disorder Episode (according to psychiatric DSM-IV criteria as determined with The Mini-International Neuropsychiatric Interview 5.0 (M.I.N.I. 5.0)
* Current (in past 6 months) use of antidepressant drugs or psychological interventions.
* History of psychosis, bipolar disorder, substance dependence or other severe, psychiatric disorder that requires specialized clinical attention. No eating disorders. This will all be measured with a brief self-report questionnaire.
* History of bariatric surgery and no current severe, life-threatening disease (assessed using self-report), and no severe cognitive impairment limiting the conduct of the study, as assessed through research staff- evaluation of feasibility of conducting the screening instruments in an adequate manner.
* Currently adhering to supervised behavioural interventions that intervene with MoodFood interventions. If persons are on specific dietary supplements that are competing with the MoodFood intervention, than persons must be willing to stop what they were using before the start of this study
* Non pregnant or breast feeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of Major depressive Disorder | 12 months
  The 12-month cumulative incidence of Major Depressive Disorder (MDD), defined according to the standard psychiatric DSM-IV criteria using The Mini-International Neuropsychiatric Interview 5.0 at 12 months

SECONDARY OUTCOMES:
Depressive Symptomatology PHQ-9 | 3, 6 and 12 months
  Depressive Symptomatology assessed with the Patient Health Questionnaire (PHQ-9) (Kroenke, Spitzer, & Williams, 2001)
Depressive symptomatology IDS30-SR | 3, 6 and 12 months
  Depressive symptomatology according the Inventory of Depressive Symptomatology (IDS30-SR) (Rush, Gullion, Basco, Jarrett, & Trivedi, 1996)
Food and eating behaviour (TEFQ-R18) | 3, 6 and 12 months
  The Three-factor Eating Questionnaire (TEFQ-R18) (Karlsson, Persson, Sjöström, & Sullivan, 2000)
Food behaviour questionnaire | 3, 6 and 12 months
  Food Behaviour Questionnaire on meal pattern, snacking behaviour, and other food-related behaviours in the past two weeks, such as mindful eating, cooking and shopping skills, etc.
Food intake GA2LEN-FFQ | 6 and 12 months
  The GA2LEN-FFQ (Garcia-Larsen et al., 2011): 6 and 12 months later
Physical activity and sedentary behavior (composite) | 3, 6 and 12 months
  Short Questionnaire to Assess Health-Enhancing Physical Activity (SQUASH) (Wendel-Vos, Schuit, Saris, & Kromhout, 2003) and The Sedentary Behavior Questionnaire (SBQ, Rosenberg et al., 2010)
Body weight perception | 3, 6 and 12 months
  The Stunkard figure rating scale (Stunkard, Sørensen, & Schulsinger, 1983)
Anxiety symptoms (GAD-7) | 3, 6 and 12 months
  Generalized Anxiety Disorder Assessment (GAD-7) (Spitzer, Kroenke, Williams, & Löwe, 2006)
Health-related quality of life | 3, 6 and 12 months
  EuroQol instrument EQ-5D-5L (EuroQol Group, 1990)
Sedentary behaviour by accelerometry in some participants | 3, 6 and 12 months
  Monitoring of sedentary and activity behaviour by accelerometry in some participants

OTHER OUTCOMES:
Body weight (composite) | 3, 6 and 12 months
  Measured height, body weight, waist and hip circumference according to standardized measurement protocols, and calculated body mass index
Body composition (composite) | 3, 6 and 12 months
  Fat mass, fat-free mass and percentage body fat will be accurately assessed using whole body air-displacement plethysmography in participants from one site.
Behavioral functionality Assessed with Behavioral activation for Depression Scale (BADS) | 3, 6 and 12 months
  Activation rumination, avoidance, work/school and social impairment. Assessed with Behavioral activation for Depression Scale (BADS) (Kanter, JW et al., 2012)
Physical activity and habits strength | 3, 6 and 12 months
  Self-Report Behavioural Automaticity Index (SRBAI) (Gardner, Abraham, Lally, & de Bruijn, 2012)
Blood sample ( blood levels of the nutrients provided with the multi-nutrient supplement) | 6 and 12 months
  In a random subsample of trial participants (n=50 per intervention arm) blood samples will be collected at baseline, and after 6 and 12 months to measure blood levels of the nutrients provided with the multi-nutrient supplement
Self-report of Somatic health status | 6 and 12 months
  Self-report of somatic/chronic diseases and family's medical history, smoking, alcohol consumption and medication/supplements use at 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Marjolein Visser, PhD, Study Director — VU University of Amsterdam
Locations (4):
- Universität Leipzig, Leipzig, Saxony, Germany
- VU Amsterdan University, Amsterdam, North Holland, Netherlands
- University of Balearic Islands, Palma de Mallorca, Balearic Islands, Spain
- University of Exeter, Exeter, Devon, United Kingdom

REFERENCES:
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Garcia-Larsen V, Luczynska M, Kowalski ML, Voutilainen H, Ahlstrom M, Haahtela T, Toskala E, Bockelbrink A, Lee HH, Vassilopoulou E, Papadopoulos NG, Ramalho R, Moreira A, Delgado L, Castel-Branco MG, Calder PC, Childs CE, Bakolis I, Hooper R, Burney PG; GA2LEN-WP 1.2 'Epidemiological and Clinical Studies'. Use of a common food frequency questionnaire (FFQ) to assess dietary patterns and their relation to allergy and asthma in Europe: pilot study of the GA2LEN FFQ. Eur J Clin Nutr. 2011 Jun;65(6):750-6. doi: 10.1038/ejcn.2011.15. Epub 2011 Mar 23. PMID 21427744
- [Background] Gardner B, Abraham C, Lally P, de Bruijn GJ. Towards parsimony in habit measurement: testing the convergent and predictive validity of an automaticity subscale of the Self-Report Habit Index. Int J Behav Nutr Phys Act. 2012 Aug 30;9:102. doi: 10.1186/1479-5868-9-102. PMID 22935297
- [Background] Kanter JW, Mulick PS, Busch AM, Berlin KS, Martell CR. (2012) . Behavioral Activation for Depression Scale (BADS) (Long and Short Form). Measurement Instrument Database for the Social Science. Retrieved from www.midss.ie
- [Background] Karlsson J, Persson LO, Sjostrom L, Sullivan M. Psychometric properties and factor structure of the Three-Factor Eating Questionnaire (TFEQ) in obese men and women. Results from the Swedish Obese Subjects (SOS) study. Int J Obes Relat Metab Disord. 2000 Dec;24(12):1715-25. doi: 10.1038/sj.ijo.0801442. PMID 11126230
- [Background] Rosenberg DE, Norman GJ, Wagner N, Patrick K, Calfas KJ, Sallis JF. Reliability and validity of the Sedentary Behavior Questionnaire (SBQ) for adults. J Phys Act Health. 2010 Nov;7(6):697-705. doi: 10.1123/jpah.7.6.697. PMID 21088299
- [Background] Rush AJ, Gullion CM, Basco MR, Jarrett RB, Trivedi MH. The Inventory of Depressive Symptomatology (IDS): psychometric properties. Psychol Med. 1996 May;26(3):477-86. doi: 10.1017/s0033291700035558. PMID 8733206
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Stunkard AJ, Sorensen T, Schulsinger F. Use of the Danish Adoption Register for the study of obesity and thinness. Res Publ Assoc Res Nerv Ment Dis. 1983;60:115-20. No abstract available. PMID 6823524
- [Background] Wendel-Vos GC, Schuit AJ, Saris WH, Kromhout D. Reproducibility and relative validity of the short questionnaire to assess health-enhancing physical activity. J Clin Epidemiol. 2003 Dec;56(12):1163-9. doi: 10.1016/s0895-4356(03)00220-8. PMID 14680666
- [Derived] Owens M, Watkins E, Bot M, Brouwer IA, Roca M, Kohls E, Penninx B, van Grootheest G, Cabout M, Hegerl U, Gili M, Visser M; MooDFOOD Prevention Trial Investigators. Acceptability and feasibility of two interventions in the MooDFOOD Trial: a food-related depression prevention randomised controlled trial in overweight adults with subsyndromal symptoms of depression. BMJ Open. 2020 Sep 15;10(9):e034025. doi: 10.1136/bmjopen-2019-034025. PMID 32933954
- [Derived] Paans NPG, Bot M, Brouwer IA, Visser M, Gili M, Roca M, Hegerl U, Kohls E, Owens M, Watkins E, Penninx BWJH; MooDFOOD Prevention Trial Investigators. Effects of food-related behavioral activation therapy on eating styles, diet quality and body weight change: Results from the MooDFOOD Randomized Clinical Trial. J Psychosom Res. 2020 Oct;137:110206. doi: 10.1016/j.jpsychores.2020.110206. Epub 2020 Jul 30. PMID 32798835
- [Derived] Baldofski S, Mauche N, Dogan-Sander E, Bot M, Brouwer IA, Paans NPG, Cabout M, Gili M, van Grootheest G, Hegerl U, Owens M, Roca M, Visser M, Watkins E, Penninx BWJH, Kohls E. Depressive Symptom Clusters in Relation to Body Weight Status: Results From Two Large European Multicenter Studies. Front Psychiatry. 2019 Nov 21;10:858. doi: 10.3389/fpsyt.2019.00858. eCollection 2019. PMID 31824355
- [Derived] Grasso AC, Olthof MR, van Dooren C, Roca M, Gili M, Visser M, Cabout M, Bot M, Penninx BWJH, van Grootheest G, Kohls E, Hegerl U, Owens M, Watkins E, Brouwer IA; MooDFOOD Prevention Trial Investigators. Effect of food-related behavioral activation therapy on food intake and the environmental impact of the diet: results from the MooDFOOD prevention trial. Eur J Nutr. 2020 Sep;59(6):2579-2591. doi: 10.1007/s00394-019-02106-1. Epub 2019 Oct 23. PMID 31642985
- [Derived] Bot M, Brouwer IA, Roca M, Kohls E, Penninx BWJH, Watkins E, van Grootheest G, Cabout M, Hegerl U, Gili M, Owens M, Visser M; MooDFOOD Prevention Trial Investigators. Effect of Multinutrient Supplementation and Food-Related Behavioral Activation Therapy on Prevention of Major Depressive Disorder Among Overweight or Obese Adults With Subsyndromal Depressive Symptoms: The MooDFOOD Randomized Clinical Trial. JAMA. 2019 Mar 5;321(9):858-868. doi: 10.1001/jama.2019.0556. PMID 30835307
- [Derived] Roca M, Kohls E, Gili M, Watkins E, Owens M, Hegerl U, van Grootheest G, Bot M, Cabout M, Brouwer IA, Visser M, Penninx BW; MooDFOOD Prevention Trial Investigators. Prevention of depression through nutritional strategies in high-risk persons: rationale and design of the MooDFOOD prevention trial. BMC Psychiatry. 2016 Jun 8;16:192. doi: 10.1186/s12888-016-0900-z. PMID 27277946